CLINICAL TRIAL: NCT05305872
Title: The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine
Brief Title: Gandouling in the Treatment of Wilson's Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jun Li (Other)
Responsible Party: Sponsor-Investigator, Jun Li, associate chief physician, The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine
Organization: The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GWPS
Record Dates: First submitted 2021-11-24; First posted 2022-03-31 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Wilson's Disease
MeSH Terms: conditions — Hepatolenticular Degeneration | interventions — gluconic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Gandouling
  Interventions: Drug: Gandouling
- Control group (Placebo Comparator): Zinc gluconate
  Interventions: Drug: Gandouling

INTERVENTIONS:
Drug: Gandouling — The experimental group was given gandouling tablet + zinc gluconate simulant; The course of treatment was 24 weeks.
  Other Names: zinc gluconate

SUMMARY:
To evaluate the efficacy and safety of gandouling tablet in the treatment of clinical symptoms of Wilson's diasease.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of gandouling tablet in the treatment of clinical symptoms of Wilson's diasease.Test various indicatorsbefore test, 4 weeks, 12 weeks and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Comply with the diagnosis of Wilson's disease "Guidelines for Diagnosis and Treatment of Wilson's disease 2021"
* The diagnosis of TCM syndromes complies with the syndrome of phlegm and blood stasis; Other copper-removing drugs
* Patients who have been treated with complexing agents for copper-removing treatment can enter the study after a 2-week washout period
* Age ≥15 years
* Informed consent of patients or legal representatives, And sign the informed consent form.

Exclusion Criteria:

* Severe cerebral WD patients: obvious torsion spasm, dysphagia, or bed rest and other severe neurological impairment will interfere with the safety of the subjects (UWDRS Part I neurological function score ≥156 points)
* Severe liver Type WD patients: Decompensated liver cirrhosis or liver cancer, manifested as portal hypertension, ascites, splenomegaly (WBC<3.0*109/L, PLT<50*1012/L), esophageal varices, gastrointestinal bleeding, Moderate to severe anemia or hepatic encephalopathy; severe liver fibrosis shown by imaging or any laboratory abnormality (UWDRS liver function score ≥ 17 points)
* Moderate to severe depression, recent suicidal thoughts or behavior, Severe psychiatric symptoms (UWDRS Part III Psychiatric Symptom Score ≥ 54 points)
* History of epileptic seizures within 6 months
* Complicated with serious diseases such as brain tumors, brain trauma, blood diseases, Cardiogenic diseases, HIV, etc.
* Nephritis, nephrotic syndrome, or kidney disease stage 3 or more
* Pregnant, planned pregnancy or breastfeeding women
* Cognitive dysfunction MMSE≤26 points
* Those who are currently participating in other clinical trials
* Cannot comply with the follow-up plan

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Unified Wilson's Disease Rating Scale(UWDRS) | Baseline, before the study
  Unified Wilson's Disease Rating Scale(UWDRS),the minimum is 0, and the maximum value is 320. Higher scores mean a worse outcome.
Unified Wilson's Disease Rating Scale(UWDRS) | 4 weeks
  Unified Wilson's Disease Rating Scale(UWDRS). Higher scores mean a worse outcome.
Unified Wilson's Disease Rating Scale(UWDRS) | 12 weeks
  Unified Wilson's Disease Rating Scale(UWDRS).Higher scores mean a worse outcome.
Unified Wilson's Disease Rating Scale(UWDRS) | 24 weeks
  Unified Wilson's Disease Rating Scale(UWDRS).Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
24-hour urinary copper | Baseline, before the study
  24-hour urinary copper.Higher scores mean a worse outcome.
24-hour urinary copper | 4 weeks
  24-hour urinary copper.Higher scores mean a worse outcome.
24-hour urinary copper | 12 weeks
  24-hour urinary copper.Higher scores mean a worse outcome.
24-hour urinary copper | 24 weeks
  24-hour urinary copper.Higher scores mean a worse outcome.
non-ceruloplasmin bound copper (NCC) | Baseline, before the study
  non-ceruloplasmin bound copper (NCC).Higher scores mean a worse outcome.
non-ceruloplasmin bound copper (NCC) | 4 weeks
  non-ceruloplasmin bound copper (NCC).Higher scores mean a worse outcome.
non-ceruloplasmin bound copper (NCC) | 12 weeks
  non-ceruloplasmin bound copper (NCC).Higher scores mean a worse outcome.
non-ceruloplasmin bound copper (NCC) | 24 weeks
  non-ceruloplasmin bound copper (NCC).Higher scores mean a worse outcome.

OTHER OUTCOMES:
Global Assessment Scale (GAS) | Baseline, before the study
  Global Assessment Scale (GAS).Higher scores mean a worse outcome.
Global Assessment Scale (GAS) | 4 weeks
  Global Assessment Scale (GAS).Higher scores mean a worse outcome.
Global Assessment Scale (GAS) | 12 weeks
  Global Assessment Scale (GAS).Higher scores mean a worse outcome.
Global Assessment Scale (GAS) | 24 weeks
  Global Assessment Scale (GAS).Higher scores mean a worse outcome.
Short Form-36 Questionnaire (SF-36) | Baseline, before the study
  Short Form-36 Questionnaire (SF-36).Higher scores mean a worse outcome.
Short Form-36 Questionnaire (SF-36) | 4 weeks
  Short Form-36 Questionnaire (SF-36).Higher scores mean a worse outcome.
Short Form-36 Questionnaire (SF-36) | 12 weeks
  Short Form-36 Questionnaire (SF-36).Higher scores mean a worse outcome.
Short Form-36 Questionnaire (SF-36) | 24 weeks
  Short Form-36 Questionnaire (SF-36).Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Jun Li, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ding Y, Cao K, Yang W, Hu S, Zhang J, Yang Y, Zhang X. Mapping neurological symptoms and muscle tension representations in impaired gray matter volume of Wilson disease. Front Neurol. 2025 Jun 5;16:1560848. doi: 10.3389/fneur.2025.1560848. eCollection 2025. PMID 40538652